CLINICAL TRIAL: NCT05844670
Title: CHildren Treated With Vincristine: A Trial Regarding Pharmacokinetics, DNA And Toxicity of Targeted Therapy In Pediatric Oncology Patients.
Acronym: CHAPATI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moi University (Other)
Collaborators: Princess Maxima Center for Pediatric Oncology (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V314092022
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Pediatric Cancer
Keywords: Pharmacokinetics; Vincristine-induced peripheral neuropathy; Pediatric oncology; Vincristine; Individualized dosing
MeSH Terms: conditions — Neoplasms | interventions — Vincristine

STUDY DESIGN:
Intervention Model Description: This will be a prospective cohort study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vincristine (Experimental): A dose advice for vincristine will be given based on vincristine concentrations in blood samples and toxicity monitoring.
  Interventions: Drug: Vincristine

INTERVENTIONS:
Drug: Vincristine — The initial vincristine dosage will be according to institutional treatment protocol. After vincristine administration, three blood samples will be taken at T=1, T=1.5 and T=4 hours. The concentration of vincristine will be analyzed in the samples. If the concentration of 2 or more samples is lower than the reference concentration and there is no toxicity, an advice will be given to increase dosage by 20%. Whether or not a dosage is given, vincristine concentrations will be measured again for the next dose administration.
  For the feasibility study, both venous blood samples and finger prick blood samples using Mitra tips will be taken. The cycle can be repeated maximum 2 times.
  For the rest of the study, finger prick blood samples using Mitra tips will be taken. The cycle can be repeated maximum 3 times.
  Toxicity will be monitored through physical exam and questionnaire, bilirubin levels and clinical status of the patient.

SUMMARY:
The goal of this clinical trial is to individualize the dosage of vincristine, a chemotherapy drug, in children with cancer. The main question it aims to answer is: can vincristine dosage be optimized while carefully monitoring toxicity.

The following will happen:

* Participants will receive vincristine according to the institutional treatment protocol.
* After receiving vincristine, blood samples will be taken at three time points.
* The amount of vincristine in the blood samples will be determined.
* If the amount of vincristine in the blood samples is lower than the reference and the participants do not experience toxicity due to vincristine, the dose of vincristine may be increased.
* Toxicity will be carefully monitored.

DETAILED DESCRIPTION:
Vincristine is among the most widely used and potentially effective chemotherapeutic agents in pediatric oncology patients. However, in black African children it may be sub optimally dosed due to genetic differences in the metabolism of vincristine. This study aims to optimize the dosing regimen of vincristine while carefully monitoring toxicity.

This will be a prospective cohort study consisting of two parts: a feasibility study and the rest of the study. In the feasibility study, 15 children aged 5-14 years who are scheduled to receive at least 2 vincristine administrations can be included. After the administration of vincristine, venous blood samples and finger prick blood samples will be taken to determine the vincristine concentrations. The samples will be shipped to and analyzed in the Netherlands to determine the vincristine concentration in each sample. Based on this, a dose advise will be given for subsequent vincristine administrations. This cycle will be repeated maximum 2 times but maximum 1 dose advice is given. Toxicity will be monitored by determination of the bilirubin, by questionnaires and by physical examination to check for signs of peripheral neuropathy. In the rest of the study, in which 85 children will be included, only finger prick samples will be taken.

ELIGIBILITY:
Feasibility study:

Inclusion Criteria:

* Black patients aged 5-14 years with a malignancy for which they are scheduled to receive a minimum of two VCR administrations as part of their treatment protocol: acute lymphoblastic leukemia, non-Hodgkin's lymphoma, rhabdomyosarcoma, neuroblastoma, nephroblastoma, retinoblastoma.
* Written informed consent

Exclusion Criteria:

* Severe malnutrition
* Total bilirubin >3 times upper limit of normal
* Pre-existent severe mental retardation e.g. Down syndrome
* Pre-existent peripheral neuropathy (CTCAE constipation, peripheral sensory neuropathy, peripheral motor neuropathy, or neuralgia ≥ 2 or ped-mTNS ≥ 5)

Rest of the study:

Inclusion Criteria:

* Black patients aged 2-14 years with a malignancy for which they are scheduled to receive a minimum of four VCR administrations as part of their treatment protocol: acute lymphoblastic leukemia, non-Hodgkin's lymphoma, rhabdomyosarcoma, neuroblastoma, nephroblastoma, retinoblastoma.
* Written informed consent

Exclusion Criteria:

* Severe malnutrition
* Total bilirubin >3 times upper limit of normal
* Pre-existent severe mental retardation e.g. Down syndrome
* Pre-existent peripheral neuropathy (CTCAE constipation, peripheral sensory neuropathy, peripheral motor neuropathy, or neuralgia ≥ 2 or ped-mTNS ≥ 5)

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Adapting vincristine dosage | Through study completion, an average of four months per patient (depending on treatment protocol).
  The number of patients in whom it is possible to adapt vincristine dosage based on vincristine concentrations in the blood at three time points and the presence of side-effects.

SECONDARY OUTCOMES:
Vincristine-induced peripheral neuropathy | Through study completion, an average of four months per patient (depending on treatment protocol).
  The number of patients who develop vincristine-induced peripheral neuropathy (VIPN) and the degree of VIPN. VIPN is measured using the CTCAE v5 items peripheral sensory neuropathy, peripheral motor neuropathy, neuralgia and constipation. In children aged 5 or above, VIPN will also be assessed with the ped-mTNS.
Genetics | Through study completion, an average of four months per patient (depending on treatment protocol).
  The association between pharmacogenomic parameters and the concentration of vincristine at three time points (T=60 minutes, T=90 minutes and T=240 minutes after vincristine administration) and vincristine-induced peripheral neuropathy using CTCAE v5 and ped-mTNS.
Vincristine pharmacokinetics | Through study completion, an average of four months per patient (depending on treatment protocol).
  The median vincristine concentrations and interquartile ranges (IQR) on three time points (T=60 minutes, T=90 minutes and T=240 minutes after vincristine administration).

CONTACTS AND LOCATIONS:
Overall Officials: Festus M Njuguna, MD, PhD, Principal Investigator — Moi University
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Rift Valley, Kenya

IPD SHARING:
Plan to Share IPD: Yes
The data are available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study protocol and ICF is already available upon request. Upon completion of the study, the SAP, CSR and analytic code will be accessible for unlimited amount of time.
Access Criteria: The data are available upon reasonable request.